CLINICAL TRIAL: NCT00286689
Title: Effects of Growth Hormone in Chronically Ill Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Record Owner no longer with the institution
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0403-239
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Hurler Syndrome; Cerebral Palsy; Juvenile Rheumatoid Arthritis; Crohn Disease; HIV Infections
MeSH Terms: conditions — Mucopolysaccharidosis I; Cerebral Palsy; Arthritis, Juvenile; Crohn Disease; HIV Infections | interventions — Growth Hormone; Absorptiometry, Photon

INTERVENTIONS:
Drug: Growth Hormone
Procedure: Whole body Protein turnover
Procedure: DEXA scan

SUMMARY:
The specific aims for this study are -

1. To determine the effect of GH on height, height velocity, body weight and lean body mass. This specific aim tests the hypothesis that GH significantly improves height, height velocity, weight, weight velocity and lean body mass in chronically ill children who have grown poorly despite adequate nutritional rehabilitation.
2. To determine the effect of GH on whole body protein turnover (WBPT), IGF-1 levels and on cytokines. This specific aim tests the hypothesis that chronically ill children have increased catabolism, caused by high levels of circulating cytokines and low levels of IGF-1, and that these abnormalities improve with GH treatment.
3. Evaluation of bone mineral density and bone turnover. This specific aim tests the hypothesis that bone density is low in chronically ill children secondary to increased osteoclast activity correlating with elevated cytokine levels.

We hypothesize that the anabolic effects of growth hormone (GH) will improve the height and weight of chronically ill children who have failed to grow despite receiving adequate nutrition via gastrostomy tube or oral supplementation.

DETAILED DESCRIPTION:
We will test our hypotheses by using a pilot study, in which we will recruit 18 chronically ill children from our clinical practice. We will obtain medical records for each patient 12 months prior to starting the study. Those patients without pre-study medical records will be studied for 12 months prior to starting GH. If we can obtain 6 months of prior medical records, then the patients will be studied for 6 months before starting GH. Anything less than 6 months will be studied for the full 12 months prior to starting GH. Patients will receive treatment with GH (0.3 mg/kg/wk) for 12 months and their growth will be compared to the year before treatment. All subjects will be followed every three months for the entire study. We will measure height and weight using a standardized stadiometer and scale, respectively, every three months during the study. From these measurements we will calculate height and weight velocity and height and weight Z score. Lean body mass (LBM) will be measured by DEXA every six months. Utilizing the stable isotope 1-[13C] leucine, we will measure whole body protein turnover (WBPT). Measurements of WBPT will be correlated with LBM and changes in height and weight velocity. This data will be compared to that from age matched normal children (archival data maintained by the PI). We will measure IGF-1 and the cytokines TNF-α, IL-6 and IL 10 at baseline and very six months. We will evaluate GH effects on these levels.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-17 years
* Tanner stages 1-3
* Each child must have received adequate nutritional therapy supplied by aggressive oral supplementation, gastrostomy tube, or TPN for at least 1 year prior to enrollment.
* All children will have been referred for continued poor growth and will be less than the 10th percentile for height compared to age and gender normal values.
* low IGF-1 level at the time of enrollment (measured in the Endocrine clinic).
* Chronic illness to be included are Hurler Syndrome (MPS-1) with short stature and muscle wasting, cerebral palsy with muscle wasting, juvenile rheumatoid arthritis with muscle wasting and short stature, Crohn's disease and HIV infection.

Exclusion Criteria:

* previous diagnosis with diabetes, chronic fevers (temp > 101.5) or chronic bacterial infection.
* substantial change in steroid dosing, or having a formerly steroid negative patient start long-term-steroids (anticipated use greater that 7 days

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-02-03 (Actual); Primary Completion 2006-02-03 (Actual); Study Completion 2006-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center of Dallas, Dallas, Texas, United States